CLINICAL TRIAL: NCT07218107
Title: Neurostimulation Exosuit Augmented Training (NEAT) in the Clinic Using a Wearable Propulsion Neuroprosthesis
Brief Title: Neurostimulation Exosuit Augmented Training (NEAT) in the Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Lou Awad, PT, DPT, PhD, Associate Professor, Physical Therapy, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 5715-FESTx
Record Dates: First submitted 2024-07-02; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: functional electrical stimulation; neuroprosthesis; gait training; chronic stroke; exosuit; neurostimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- NEAT Program (Experimental): Neurostimulation Exosuit Augmented Training (NEAT) refers to gait training with electrical stimulation exosuits, sometimes known as neuroprostheses. NEAT incorporates a speed-based approach that asks participants to walk at fast speeds on the treadmill and overground. Goal-directed walking practice if facilitated by a physical therapist who provides cues and feedback emphasizing a focus on increasing walking speed and forward propulsion. Training is progressively challenging based on environmental complexity and practice variability. NEAT includes 12 training sessions administered 2-3 times per week. Each session includes 30 minutes of gait training.
  Interventions: Device: Neurostimulation Exosuit

INTERVENTIONS:
Device: Neurostimulation Exosuit — A neurostimulation exosuit (i.e., neuroprosthesis) is a textile-based device worn on the paretic lower limb. Neuroprostheses deliver functional electrical stimulation through non-invasive surface electrodes placed on the front and the back of the leg, providing swing-phase dorsiflexor assistance for foot clearance and stance-phase plantarflexor assistance for forward propulsion, respectively. Neurostimulation assistance is provided synchronously with the wearer's gait, based on inertial sensors in the shoes that measure the wearer's unique walking pattern.
  Other Names: Neuroprosthesis

SUMMARY:
The primary goal of this study is to understand the feasibility and rehabilitative effects of a Neurostimulation Exosuit Augmented Training (NEAT) program designed to provide high-intensity gait training in progressively challenging environments for individuals in the chronic phase of stroke recovery. The investigators will monitor feasibility of the training program and assess walking endurance and energy efficiency before and after the training to quantify effects of the training program on the recovery of walking function driven by improvements in forward propulsion and symmetry between limbs. Participants will complete pre-training and post-training evaluations alongside 12 gait training sessions across 4-5 weeks.

DETAILED DESCRIPTION:
Functional electrical stimulation (FES) is commonly used to manage foot drop in people with post-stroke hemiparesis. Emerging use of FES applied to the paretic plantarflexors to facilitate push-off ability during walking has been limited to the treadmill and highly supervised laboratory-based settings. This novel neurostimulation exosuit (i.e., neuroprosthesis) enables overground gait training in environments of varying complexity by giving clinicians the ability to modulate neurostimulation timing and intensity delivered to the dorsiflexors for swing-phase foot clearance and to the plantarflexors for stance-phase plantarflexor forward propulsion. Combined with progressive, high-intensity, task-specific gait training, as has been performed previously with soft robotic exosuits developed by the same research group, this propulsion neuroprosthesis will leverage i) immediate gait assistance from the neurostimulation to facilitate high intensity training without sacrificing gait quality and ii) neurorestorative properties of FES to encourage the recovery motor function to affected muscles.

The primary objective of this study seeks to understand the feasibility and rehabilitative effects of a Neurostimulation Exosuit Augmented Training (NEAT) program designed to provide high-intensity speed-driven gait training in progressively challenging environments. The investigators hypothesize that the NEAT program will safely provide a standard dose of gait rehabilitation training within a clinic setting and that the training will result in clinically meaningful gains in walking endurance and energy efficiency driven by improvements in forward propulsion and symmetry between limbs.

Secondary objectives of this study seek to assess the effects of the NEAT program on neuromuscular control to the paretic plantarflexors (i.e., central drive). The investigators hypothesize that repeated training with neurostimulation to the dorsiflexors and plantarflexors will result in increased neuromuscular control to the paretic plantarflexors.

The NEAT program will consist of 14 total study visits: i) Pre-training Evaluation, ii) NEAT Training (12 sessions, 2-3 times per week), iii) Post-training Evaluation. The neurostimulation exosuit used in this study was developed for investigational use only by investigators at the Boston University Neuromotor Recovery Laboratory, the Harvard University BioDesign Lab, and the Harvard University Move Lab.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years old
* History of stroke event occurring at least 6 months ago
* Observable gait deficits characteristic of post-stroke hemiparesis
* Independent ambulation for at least 30 meters (with an assistive device if needed but without a rigid brace for the ankle)
* Ankle dorsiflexion range of motion at least to neutral (i.e., 90 degrees between the shank and the foot)
* Resting heart rate between 40 - 100 bpm (inclusive)
* Resting blood pressure between 90/60 and 170/90 mmHg (inclusive)
* HIPAA authorization to allow communication with healthcare provider as needed during the study period
* Medical clearance by a physician

Exclusion Criteria:

* NIH Stroke Scale Question 1b score > 1 and Question 1c score > 0
* Inability to communicate with investigators
* Visual neglect or hemianopia
* History of cerebellar stroke
* Actively receiving physical therapy for walking
* More than 2 unexplained falls in the previous month
* Pressure ulcers or skin wounds located near human-device interface sites
* Pacemakers or similar electrical implants that could be affected by electrical stimulation
* Metal implants directly under the stimulation sites
* Skin allergy or other condition sensitive to the adhesive from transcutaneous neurostimulation electrode pads
* Other medical, orthopedic, and neurological conditions that prevent full participation in the research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test (6MWT) Distance | Pre-training Evaluation (baseline)
  This is a clinical test of long-distance walking function. The participant walks as far as they can safely in 6 minutes. Total distance covered in 6 minutes is the primary outcome from this test. This test will be performed without a neuroprosthesis (unassisted) and with electrical stimulation assistance from a neuroprosthesis (assisted).
Six Minute Walk Test (6MWT) Distance | Post-training Evaluation (average of 5 weeks)
  This is a clinical test of long-distance walking function. The participant walks as far as they can safely in 6 minutes. Total distance covered in 6 minutes is the primary outcome from this test. This test will be performed without a neuroprosthesis (unassisted) and with electrical stimulation assistance from a neuroprosthesis (assisted).
Six Minute Walk Test (6MWT) Speed | Pre-training Evaluation (baseline)
  Walking speed is also monitored during the 6MWT at each reference length completed (e.g., 30-meter stretch before turning around). Speed is calculated as the reference length divided by the time it took to walk that distance in meters per second (m/s). This metric will be measured during the 6MWT performed without a neuroprosthesis (unassisted) and with electrical stimulation assistance from a neuroprosthesis (assisted).
Six Minute Walk Test (6MWT) Speed | Post-training Evaluation (average of 5 weeks)
  Walking speed is assessed during the 6MWT at each reference length completed (e.g., 30-meter stretch before turning around). Speed is calculated as the reference length divided by the time it took to walk that distance in meters per second (m/s). This metric is assessed during the 6MWT performed without a neuroprosthesis (unassisted) and with electrical stimulation assistance from a neuroprosthesis (assisted).
Energy Expenditure | Pre-training Evaluation (baseline)
  Energy expenditure assessed using indirect calorimetry (COSMED K5) and is calculated as the volume of oxygen inhaled normalized by bodyweight and distance (mL O2/kg/m). This metric will be measured during the 6MWT performed without a neuroprosthesis (unassisted) and with electrical stimulation assistance from a neuroprosthesis (assisted).
Energy Expenditure | Post-training Evaluation (average of 5 weeks)
  Energy expenditure assessed using indirect calorimetry (COSMED K5) and is calculated as the volume of oxygen inhaled normalized by bodyweight and distance (mL O2/kg/m). This metric will be measured during the 6MWT performed without a neuroprosthesis (unassisted) and with electrical stimulation assistance from a neuroprosthesis (assisted).
Ten Meter Walk Test (10mWT) Speed | Pre-training Evaluation (baseline)
  This is a clinical test of short-distance walking function. The participant walks at a comfortable walking speed (CWS) and fast walking speed (FWS) on a 10-meter straight walkway. The middle six meters are used to assess speed across 3 trials for CWS and 3 trials for FWS.
Ten Meter Walk Test (10mWT) Speed | Post-training Evaluation (average of 5 weeks)
  This is a clinical test of short-distance walking function. The participant walks at a comfortable walking speed (CWS) and fast walking speed (FWS) on a 10-meter straight walkway. The middle six meters are used to assess speed across 3 trials for CWS and 3 trials for FWS.
Plantarflexor Central Drive | Pre-training Evaluation (baseline)
  Central drive is a measure of voluntary control of a muscle. The participant uses their plantarflexors to push into a torque-sensing plate. Upon reaching the plateau of a maximum voluntary contraction (MVC), a burst of electrical stimulation is delivered using the burst superimposition technique to activate any remaining muscle fibers that are not activated volitionally, obtaining the maximum force-generating ability (MFGA). Central drive is calculated as the ratio of MVC to MFGA as a percentage (i.e., 100% central drive indicates full voluntary control of the muscle). Paretic plantarflexor central drive is assessed every 3-4 training days.
Plantarflexor Central Drive | Training Day 3
  Central drive is a measure of voluntary control of a muscle. The participant uses their plantarflexors to push into a torque-sensing plate. Upon reaching the plateau of a maximum voluntary contraction (MVC), a burst of electrical stimulation is delivered using the burst superimposition technique to activate any remaining muscle fibers that are not activated volitionally, obtaining the maximum force-generating ability (MFGA). Central drive is calculated as the ratio of MVC to MFGA as a percentage (i.e., 100% central drive indicates full voluntary control of the muscle). Paretic plantarflexor central drive is assessed every 3-4 training days.
Plantarflexor Central Drive | Training Day 6
  Central drive is a measure of voluntary control of a muscle. The participant uses their plantarflexors to push into a torque-sensing plate. Upon reaching the plateau of a maximum voluntary contraction (MVC), a burst of electrical stimulation is delivered using the burst superimposition technique to activate any remaining muscle fibers that are not activated volitionally, obtaining the maximum force-generating ability (MFGA). Central drive is calculated as the ratio of MVC to MFGA as a percentage (i.e., 100% central drive indicates full voluntary control of the muscle). Paretic plantarflexor central drive is assessed every 3-4 training days.
Plantarflexor Central Drive | Training Day 9
  Central drive is a measure of voluntary control of a muscle. The participant uses their plantarflexors to push into a torque-sensing plate. Upon reaching the plateau of a maximum voluntary contraction (MVC), a burst of electrical stimulation is delivered using the burst superimposition technique to activate any remaining muscle fibers that are not activated volitionally, obtaining the maximum force-generating ability (MFGA). Central drive is calculated as the ratio of MVC to MFGA as a percentage (i.e., 100% central drive indicates full voluntary control of the muscle). Paretic plantarflexor central drive is assessed every 3-4 training days.
Plantarflexor Central Drive | Post-training Evaluation (average of 5 weeks)
  Central drive is a measure of voluntary control of a muscle. The participant uses their plantarflexors to push into a torque-sensing plate. Upon reaching the plateau of a maximum voluntary contraction (MVC), a burst of electrical stimulation is delivered using the burst superimposition technique to activate any remaining muscle fibers that are not activated volitionally, obtaining the maximum force-generating ability (MFGA). Central drive is calculated as the ratio of MVC to MFGA as a percentage (i.e., 100% central drive indicates full voluntary control of the muscle). Paretic plantarflexor central drive is assessed every 3-4 training days.
Gait Propulsion | Pre-training Evaluation (baseline)
  Propulsion is the anterior component of the ground reaction force corresponding to the push-off subtask of walking that propels a forward into the next step. Gait propulsion is assessed during the 6MWT using floor-embedded forceplates.
Gait Propulsion | Post-training Evaluation (average of 5 weeks)
  Propulsion is the anterior component of the ground reaction force corresponding to the push-off subtask of walking that propels a forward into the next step. Gait propulsion is assessed during the 6MWT using floor-embedded forceplates.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | First Training Day (Day 1)
  This is a self-report measure of usability of a device. The assessment asks about complexity of the device, need for technical support, confidence in using the device, etc. Each of the 10 questions is rated from 1 (strongly disagree) to 5 (strongly agree) and scaled with a maximum score of 100.
System Usability Scale (SUS) | Mid-Training (Day 7)
  This is a self-report measure of usability of a device. The assessment asks about complexity of the device, need for technical support, confidence in using the device, etc. Each of the 10 questions is rated from 1 (strongly disagree) to 5 (strongly agree) and scaled with a maximum score of 100.
System Usability Scale (SUS) | Last Training Day (Day 12)
  This is a self-report measure of usability of a device. The assessment asks about complexity of the device, need for technical support, confidence in using the device, etc. Each of the 10 questions is rated from 1 (strongly disagree) to 5 (strongly agree) and scaled with a maximum score of 100.
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) - Modified | First Training Day (Day 1)
  This is a self-report measure of satisfaction with an assistive device. The assessment asks about various aspects of the device, such as size, weight, comfort, etc. The questions are rated from 1 (not satisfied at all) to 5 (very satisfied). This measure has been modified by the investigators to assess only the 8 questions related to device characteristics (i.e., removed questions related to technology services).
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) - Modified | Mid-Training (Day 7)
  This is a self-report measure of satisfaction with an assistive device. The assessment asks about various aspects of the device, such as size, weight, comfort, etc. The questions are rated from 1 (not satisfied at all) to 5 (very satisfied). This measure has been modified by the investigators to assess only the 8 questions related to device characteristics (i.e., removed questions related to technology services).
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) - Modified | Last Training Day (Day 12)
  This is a self-report measure of satisfaction with an assistive device. The assessment asks about various aspects of the device, such as size, weight, comfort, etc. The questions are rated from 1 (not satisfied at all) to 5 (very satisfied). This measure has been modified by the investigators to assess only the 8 questions related to device characteristics (i.e., removed questions related to technology services).

OTHER OUTCOMES:
Functional Gait Assessment (FGA) | Pre-training Evaluation (baseline)
  This is a clinical test of stability during walking, including tasks such as walking with speed changes or head turns, stepping over obstacles, walking backwards, and walking with eyes closed. Each of the 10 questions are scored from 0 (severe impairment) to 3 (normal) with a maximum score of 30 points.
Fugl-Meyer Assessment Lower Extremity Subsection (FMLE) | Pre-training Evaluation (baseline)
  This is a clinical test of motor recovery from hemiplegic stroke. Each task is scored from 0 (cannot perform) to 2 (performs fully) with a maximum score of 34 points.
Physical Activity Scale for the Elderly (PASE) - Modified | Pre-training Evaluation (baseline)
  This is a self-report measure of physical activity level used to assess the effectiveness of exercise interventions. The assessment asks how often in the past week a person participates in various leisure time activities, household activities, and work-related activities. The assessment is scored using calculated weights and frequency values for each of the 12 types of activity. This measure has been modified by the investigators to assess amount and frequency of physical activity "in general per week" instead of "during the past 7 days".
Activities-Specific Balance Confidence (ABC) | Pre-training Evaluation (baseline)
  This is a self-report measure of balance confidence while performing various tasks, such as walking around the house, picking up items from the floor, walking in a crowded mall, etc. Each of the 16 questions is rated on a 10-point scale from 0% (no confidence) to 100% (completely confident) with a maximum score of 100.
Timed Up and Go (TUG) | Pre-training Evaluation (baseline)
  This is a clinical test of balance, walking ability, and fall risk. The test consists of standing from a chair, walking 3 meters, turning around, walking back to the chair, and sitting in the chair, assessed across 3 trials.
Timed Up and Go (TUG) | Post-training Evaluation (average of 5 weeks)
  This is a clinical test of balance, walking ability, and fall risk. The test consists of standing from a chair, walking 3 meters, turning around, walking back to the chair, and sitting in the chair, assessed across 3 trials.
Self-Efficacy for Exercise (SEE) | Pre-training Evaluation (baseline)
  This is a self-report measure of exercise self-efficacy assessing confidence in the ability to exercise three times per week for 20 minutes under various conditions, such if a person is bored, in pain, busy, stressed, etc. Each of 9 questions is rated from 0 (not confident) to 10 (very confident) with a maximum score of 90.
Self-Efficacy for Exercise (SEE) | Post-training Evaluation (average of 5 weeks)
  This is a self-report measure of exercise self-efficacy assessing confidence in the ability to exercise three times per week for 20 minutes under various conditions, such if a person is bored, in pain, busy, stressed, etc. Each of 9 questions is rated from 0 (not confident) to 10 (very confident) with a maximum score of 90.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Awad, PT, PhD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Center for Neurorehabilitation, Boston, Massachusetts
  - Neuromotor Recovery Laboratory, Boston, Massachusetts

REFERENCES:
- [Background] Nadeau S, Gravel D, Arsenault AB, Bourbonnais D. Plantarflexor weakness as a limiting factor of gait speed in stroke subjects and the compensating role of hip flexors. Clin Biomech (Bristol). 1999 Feb;14(2):125-35. doi: 10.1016/s0268-0033(98)00062-x. PMID 10619100
- [Background] Takahashi KZ, Lewek MD, Sawicki GS. A neuromechanics-based powered ankle exoskeleton to assist walking post-stroke: a feasibility study. J Neuroeng Rehabil. 2015 Feb 25;12:23. doi: 10.1186/s12984-015-0015-7. PMID 25889283
- [Background] Bowden MG, Woodbury ML, Duncan PW. Promoting neuroplasticity and recovery after stroke: future directions for rehabilitation clinical trials. Curr Opin Neurol. 2013 Feb;26(1):37-42. doi: 10.1097/WCO.0b013e32835c5ba0. PMID 23254556
- [Background] Allen JL, Ting LH, Kesar TM. Gait Rehabilitation Using Functional Electrical Stimulation Induces Changes in Ankle Muscle Coordination in Stroke Survivors: A Preliminary Study. Front Neurol. 2018 Dec 20;9:1127. doi: 10.3389/fneur.2018.01127. eCollection 2018. PMID 30619077
- [Background] Kesar TM, Reisman DS, Higginson JS, Awad LN, Binder-Macleod SA. Changes in Post-Stroke Gait Biomechanics Induced by One Session of Gait Training. Phys Med Rehabil Int. 2015;2(10):1072. Epub 2015 Dec 28. PMID 27819067
- [Background] Awad LN, Reisman DS, Pohlig RT, Binder-Macleod SA. Identifying candidates for targeted gait rehabilitation after stroke: better prediction through biomechanics-informed characterization. J Neuroeng Rehabil. 2016 Sep 23;13(1):84. doi: 10.1186/s12984-016-0188-8. PMID 27663199
- [Background] Kesar TM, Perumal R, Reisman DS, Jancosko A, Rudolph KS, Higginson JS, Binder-Macleod SA. Functional electrical stimulation of ankle plantarflexor and dorsiflexor muscles: effects on poststroke gait. Stroke. 2009 Dec;40(12):3821-7. doi: 10.1161/STROKEAHA.109.560375. Epub 2009 Oct 15. PMID 19834018
- [Background] Palmer JA, Hsiao H, Wright T, Binder-Macleod SA. Single Session of Functional Electrical Stimulation-Assisted Walking Produces Corticomotor Symmetry Changes Related to Changes in Poststroke Walking Mechanics. Phys Ther. 2017 May 1;97(5):550-560. doi: 10.1093/ptj/pzx008. PMID 28339828
- [Background] Awad LN, Hsiao H, Binder-Macleod SA. Central Drive to the Paretic Ankle Plantarflexors Affects the Relationship Between Propulsion and Walking Speed After Stroke. J Neurol Phys Ther. 2020 Jan;44(1):42-48. doi: 10.1097/NPT.0000000000000299. PMID 31834220
- [Background] Porciuncula F, Baker TC, Arumukhom Revi D, Bae J, Sloutsky R, Ellis TD, Walsh CJ, Awad LN. Targeting Paretic Propulsion and Walking Speed With a Soft Robotic Exosuit: A Consideration-of-Concept Trial. Front Neurorobot. 2021 Jul 28;15:689577. doi: 10.3389/fnbot.2021.689577. eCollection 2021. PMID 34393750
- [Background] Awad LN, Reisman DS, Kesar TM, Binder-Macleod SA. Targeting paretic propulsion to improve poststroke walking function: a preliminary study. Arch Phys Med Rehabil. 2014 May;95(5):840-8. doi: 10.1016/j.apmr.2013.12.012. Epub 2013 Dec 28. PMID 24378803
- [Background] Sabut SK, Lenka PK, Kumar R, Mahadevappa M. Effect of functional electrical stimulation on the effort and walking speed, surface electromyography activity, and metabolic responses in stroke subjects. J Electromyogr Kinesiol. 2010 Dec;20(6):1170-7. doi: 10.1016/j.jelekin.2010.07.003. Epub 2010 Aug 6. PMID 20692180
- [Background] Kesar TM, Reisman DS, Perumal R, Jancosko AM, Higginson JS, Rudolph KS, Binder-Macleod SA. Combined effects of fast treadmill walking and functional electrical stimulation on post-stroke gait. Gait Posture. 2011 Feb;33(2):309-13. doi: 10.1016/j.gaitpost.2010.11.019. Epub 2010 Dec 22. PMID 21183351
- [Background] Collimore AN, Alvarez JT, Sherman DA, Gerez LF, Barrow N, Choe DK, Binder-Macleod S, Walsh CJ, Awad LN. A Portable, Neurostimulation-Integrated, Force Measurement Platform for the Clinical Assessment of Plantarflexor Central Drive. Bioengineering (Basel). 2024 Jan 30;11(2):137. doi: 10.3390/bioengineering11020137. PMID 38391623